CLINICAL TRIAL: NCT06633887
Title: Feasibility Evaluation of Sleep Apnea Screening with Photoplethysmography
Brief Title: TipTraQ Home Sleep Test Study, SHH
Status: Completed | Type: Observational
Sponsor: PranaQ Pte. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: TipTraQ developement SHH; N202303101 (Other: TMU-Joint Institutional Review Board)
Record Dates: First submitted 2024-10-02; First posted 2024-10-09 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy or people who has indication to conduct polysomnography (PSG).

SUMMARY:
The clinical study aims to develop and validate the TipTraQ system, created by PranaQ, a home sleep test for sleep apnea screening. The system comprises a wearable device and a cloud-based AI for estimating Total Sleep Time (TST) and Apnea-Hypopnea Index (AHI).

DETAILED DESCRIPTION:
Sleep-disordered breathing is a common disease that affects life function and quality of life, and it also imposes a great burden on the public health system. Obstructive sleep apnea accounts for the largest proportion of sleep-disordered breathing, and because of the oriental facial structure, the prevalence of sleep-disordered breathing is relatively high. The current gold standard for diagnosis OSA is polysomnography (PSG). Although the physiological information collected by PSG is complete and detailed, it requires a considerable amount of manpower and medical resources, and changes in the sleep environment also cause bias in the accuracy of inspection. So far, the tools for simple and accurate screening and diagnosis OSA are relatively limited. In this study, TipTraQ, a wearable device developed by PranaQ, was used to collect photoplethysmography (PPG) of patients during the night of PSG inspection. The reliability and validity analysis was carried out by comparing with the corresponding indicators of PSG, and the feasibility of TipTraQ as a tool for home sleep test (HST).

ELIGIBILITY:
Inclusion Criteria:

Subjects from the age of 20 and older that have an indication for an in-lab PSG study.

Exclusion Criteria:

* Heart transplant
* Heart failure, New Youk Heart Association (NYHA) classification III or IV
* Chronic opioid medication user
* Devastating severe strokes, with the modified Rankin score (mRS)≥4
* Tracheostomy
* Incapable of comprehending and signing the informed consent and questionnaires, including but not limited to subjects with severe Alzheimer's, unconscious by head trauma, or of someone with limited mental capacity
* Cannot correctly follow the order to use the TipTraQ device

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy or people who has indication to conduct polysomnography (PSG).
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index(AHI) | From the start of a single polysomnography study to the end of the recording, 1 night.
  The combined average number of apneas and hypopneas that occur per hour of sleep
Oxygen Desaturation Index(ODI) | From the start of a single polysomnography study to the end of the recording, 1 night.
  Average desaturation episodes with a decrease in the oxygen saturation of ≥4% or 3% per hour
Total Sleep Time(TST) | From the start of a single polysomnography study to the end of the recording, 1 night.
  Total sleep time during the polysomnography (PSG)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, New Taipei City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen KW, Tseng CH, Lee HC, Liu WT, Chou KT, Wu HT. Validation of a fingertip home sleep apnea testing system using deep learning AI and a temporal event localization analysis. Sleep. 2025 May 12;48(5):zsae317. doi: 10.1093/sleep/zsae317. PMID 39821673